CLINICAL TRIAL: NCT04788316
Title: A Technology-based Intervention to Reduce Alcohol Use After Bariatric Surgery
Brief Title: Reducing Alcohol Use Post-Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Lisa Matero, Assistant Scientist, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RAPS; R34AA027775 (NIH)
Record Dates: First submitted 2021-03-03; First posted 2021-03-09 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Bariatric Surgery Candidate; Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): A computerized brief intervention (CBI) followed by six months of personalized text messaging
  Interventions: Behavioral: CBI and Text messaging
- Control (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: CBI and Text messaging — A computerized brief intervention (2 sessions) followed by six months of personalized text messaging
  Arms: Intervention

SUMMARY:
Despite bariatric surgery being the most effective weight loss intervention for patients who are severely obese, as many as 1 in 5 patients will develop an alcohol use disorder after their surgery. Changes in metabolism, hormone levels, and behavior as a result of bariatric surgery alter the rewarding effects of alcohol while concurrently changing its absorption rate, putting patients at significantly elevated risk of hazardous drinking. Simply providing education to this vulnerable patient population about post-surgical risks has not been sufficient to reduce alcohol use, yet comprehensive in-person interventions are met with significant challenges, including hours-long distances between patients and their bariatric surgery programs. Thus, the long-term goal is to increase access to an empirically-supported intervention for reducing alcohol use among patients who undergo bariatric surgery by leveraging technology. This intervention, rooted in motivational interviewing and the transtheoretical model, is a two-session computerized brief intervention CBI, supplemented by six months of tailored text messaging based on participants CBI results and subsequent fluctuations in their readiness to change. The purpose of the proposed study is to optimize this technology-based intervention for patients who undergo bariatric surgery and to examine feasibility and acceptability of the intervention. In the first phase, patient interviews will be utilized to identify preferences for intervention content and treatment delivery. Ten patients will then participate in an open trial of the intervention, which will be subsequently revised based on feedback from these patients. In Phase 2, patients will be recruited between 3 and 6 months following bariatric surgery and randomized to the intervention or treatment as usual control group. All patients will complete baseline questionnaires and at 1, 3, 6, and 9 month post-assessments. The investigators expect that this intervention will be both feasible and acceptable to patients. Results will be used as preliminary data to inform a large, fully-powered clinical trial to test the larger efficacy of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Underwent a bariatric surgery procedure between 3 and 6 months prior to the recruitment date
* Has not consumed alcohol since undergoing bariatric surgery

Exclusion Criteria:

* History of an alcohol use disorder
* Never consumed alcohol prior to surgery
* Does not have a cellular phone that can receive and send text messages
* No access to internet to complete the computerized brief intervention (CBI)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Time to alcohol use | 6 months post-baseline
  The number of days that elapsed from surgery until the first alcoholic drink
Number of drinking days | 6 months post-baseline
  The number of drinking days/days abstinent
Drinks per day | 6 months post-baseline
  Average drinks per sitting

SECONDARY OUTCOMES:
Risky alcohol use | 6 months post-baseline
  Definition of at-risk drinking from the National Institute of on Alcohol Abuse and Alcoholism (i.e., more than 3 drinks in a day for women or 4 for men or more than 7 drinks in a week for women or 14 drinks for men)
Hazardous alcohol use | 6 months post-baseline
  Scores on Alcohol Use Disorder Identification Test-Concise. Scores range from 0-12, with higher scores indicating greater potential for hazardous use. Scores of 3+ for women or 4+ for men indicate hazardous use.
Importance of and confidence in the ability to abstain from alcohol | 6 months post-baseline
  Measured on 0-10 scales; with higher scores indicating greater importance and confidence

OTHER OUTCOMES:
Drinking Motives | 6 months post-baseline
  The Drinking Motives Questionnaire-Revised (DMQ-R) assesses respondents' reasons for drinking across four categories: conformity, coping, enhancement, and social. Each subscale has scores that range from 5-25, with higher scores indicating greater motivation to use alcohol.
Depression | 6 months post-baseline
  Patient Health Questionnaire depression scale (PHQ-8) will measure depression scores. Scores range from 0-24 with higher scores indicating greater levels of depression.
Anxiety | 6 months post-baseline
  Measured by the Generalized Anxiety Disorder-7 (GAD-7). Scores range from 0-21 with higher scores indicating greater levels of anxiety.
Food addiction | Baseline and 1, 3, and 9 month follow ups
  Yale Food Addiction Scale 2.0 (YFAS 2.0) will assess for symptoms of food addiction (similar to substance use disorder criteria in the DSM-V). Responses result in a symptom count that can range from 0-11 symptoms, with a higher number indicating more symptoms of food addiction. The scale can also indicate whether the symptoms are clinically significant (i.e., yes or no), and the scale can also give a determination of whether someone meets criteria for food addiction (yes or no), and if so, will determine if the addiction is considered mild, moderate, or severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller-Matero LR, Pappas C, Christopher B, Grossi R, Vanderziel A, Barnett NP, Moore RS, Bendit S, Hamann A, Carlin AM, Varban OA, Braciszewski JM. A Need for Strategies to Reduce Alcohol Use After Metabolic and Bariatric Surgery: Technology-Based Intervention and Study Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2026 Jan 7;15:e80068. doi: 10.2196/80068. PMID 41499161